CLINICAL TRIAL: NCT06468956
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled Phase III Clinical Study to Evaluate the Efficacy and Safety of SHR-1819 Injection in Patients With Moderate to Severe Atopic Dermatitis
Brief Title: Efficacy and Safety Study of SHR-1819 Injection in Adult Patients With Severe Atopic Dermatitis
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Guangdong Hengrui Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR-1819-301
Record Dates: First submitted 2024-05-24; First posted 2024-06-21 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Moderate to Severe Atopic Dermatitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SHR-1819 injection dose 1 (Experimental)
  Interventions: Drug: SHR-1819
- SHR-1819 injection dose 2 (Experimental)
  Interventions: Drug: SHR-1819
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SHR-1819 — SHR-1819 injection
  Arms: SHR-1819 injection dose 1; SHR-1819 injection dose 2
Drug: Placebo — placebo
  Arms: placebo

SUMMARY:
This trial was designed to evaluate the efficacy and safety of SHR-1819 injection in patients with atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects voluntarily sign informed consent forms prior to the commencement of any proceedings related to the study, are able to communicate smoothly with the investigator, understand and are willing to complete the study in strict compliance with the requirements of this clinical research protocol；
2. The age was ≥18 at the time of signing the informed consent and gender is unlimited;
3. Atopic dermatitis at screening (according to the 2014 American Society of Dermatology guideline criteria, see Annex 1) and disease duration for at least 1 year before screening as judged by the investigator;
4. EASI ≥ 16, IGA ≥ 3, BSA ≥ 10% during the screening and baseline periods;
5. TCS was not optimal or not tolerated by the investigator.

Exclusion Criteria:

1. Pregnant or lactating women;
2. Major surgeries are planned for the duration of the study;
3. History of previous atopic corneal conjunctivitis involving the cornea;
4. History of clinically significant diseases (e.g., circulatory system abnormalities, endocrine system abnormalities, neurological disorders, hematologic disorders, immune system disorders, psychiatric disorders, and metabolic instability) that the researcher believes that participation in the study poses a risk to the safety of the subject or that the disease/illness worsens during the study period will affect the effectiveness or safety analysis;
5. Subjects have had or are currently clinically significant diseases or abnormalities;
6. Screening for people with a history of heavy alcohol consumption or substance abuse in the 3 months prior to screening;
7. The drug has been used in the previous 6 months;
8. Screening of subjects with malignancy within the first 5 years (except completely cured cervical cancer in situ and non-metastatic cutaneous squamous cell carcinoma or basal cell carcinoma);
9. Other comorbid (or co-occurring) skin disorders may be affected in the study evaluation;
10. Any cause that the researchers believe would prevent the participants from participating in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 652 (Actual)
Dates: Start 2024-06-14 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
At 16 weeks, the proportion of subjects who achieved eczema area and severity index (EASI) -75 (EASI score decreased ≥75% from baseline) | up to 16 weeks
  The extent of area is assessed using the EASI scale
At week 16, the proportion of participants with an overall investigator assessment (IGA) score of 0 or 1 and a decrease of ≥2 points from baseline | up to 16 week
  The overall degree of improvement was assessed using the IGA scale

SECONDARY OUTCOMES:
The proportion of subjects whose weekly mean of the daily (PP-NRS) score decreased by 4 points from baseline at Week 16 | up to 16 weeks
  Prtch improvement was assessed using the pruritus scale
At week 16, the proportion of subjects who achieved EASI-90 (EASI score ≥90% lower than baseline) | up to 16 weeks
  The extent of area is assessed using the EASI scale
Proportion of subjects reaching EASI-75 at other visit viewpoints | up to 52 weeks
  The extent of area is assessed using the EASI scale
The proportion of subjects with IGA score of 0 or 1 and 2 points from baseline | up to 52 weeks
  The overall degree of improvement was assessed using the IGA scale
Proproportion of subjects with a 2 points from baseline at each iGA | up to 52 weeks
  The overall degree of improvement was assessed using the IGA scale
Percentage of change and change from baseline in EASI per visit viewpoint | up to 52 weeks
  The extent of area is assessed using the EASI scale
Percentage of subjects with weekly mean PP-NRS scores of 3 points from baseline | up to 52 weeks
  Prtch improvement was assessed using the pruritus scale
Percentage of change and change from baseline in the Skin Quality of Life Index Questionnaire (DLQI) score at each visit viewpoint | From the beginning of administration to the 52 week
  Subject quality of life was assessed using the DLQI scale
Percentage of change from baseline in eczema self-assessment (POEM) scores at each viewpoint | From the beginning of administration to the 52 week
  Subject quality of life was assessed using the POEM scale
The time of SHR-1819 in the serum | From the beginning of administration to the 52th week
  The concentration of SHR-1819 in plasma will be determined
The concentration of SHR-1819 in serum: AUC | From the beginning of administration to the 52th week
  The concentration of SHR-1819 in plasma will be determined
Changes in the level of IgE in the serum | From the beginning of administration to the 52th week
  Changes in the level of biomarkers in serum

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Fudan University HuaShan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided